CLINICAL TRIAL: NCT06275542
Title: Ability to Maintain Saturation Levels Without Oxygen Supplementation as a Extubation Criterion Without TOF Monitoring Equipment
Brief Title: Ability to Maintain Saturation Levels Without Oxygen Supplementation as a Extubation Criteria Without TOF Monitoring Equipment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surabaya (Other)
Collaborators: Anesthesiology and Intensive Therapy, Faculty of Medicine, Universitas Gadjah Mada (Unknown)
Responsible Party: Principal Investigator, Ardyan Prima Wardhana, Ardyan Prima Wardhana, MD, University of Surabaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USurabaya
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia Intubation Complication
Keywords: Extubation; residual paralysis; Quantitative TOF monitoring; reversal
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Intervention Model Description: The study was conducted through a randomized clinical trial with blinding of observers. Two parallel groups were selected to compare the incidence of paralysis in the recovery room. The research samples were collected using non-probability sampling method through consecutive enrollment over a specific period. This study consisted of 3 comparisons distinguished based on the type of volatile anesthetic gas maintenance and neuromuscular blockade agent, namely:
  * Comparison 1: The volatile anesthetic gas used was sevoflurane and the muscular blockade agent used was rocuronium.
  * Comparison 2: The volatile anesthetic gas used was isoflurane and the muscular blockade agent used was rocuronium.
  * Comparison 3: The volatile anesthetic gas used was sevoflurane and the muscular blockade agent used was atracurium.
Who Masked: Participant, Outcomes Assessor
Masking Description: Upon arrival in the recovery room, all subjects were fitted with SpO2, EKG, NIBP monitors, and the TOF monitoring device. TOF values were measured by a second researcher who was unaware of the type of intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical extubation strategy without TOF monitoring (Experimental): Extubation without TOF monitoring strategy: the administration of neostigmine reversal with a dose based on the degree of blockade without TOF monitoring, and extubation is performed at least 15 minutes after reversal if the patient can maintain SpO2 > 95% for 3 minutes after receiving room air without oxygen supplementation.
  Interventions: Drug: Neostigmine; Procedure: Air chalenge prior to extubation; Device: Train of Four monitoring device in recovery room
- Clinical extubation strategy with TOF monitoring (Active Comparator): Extubation with quantitative TOF monitoring strategy: neostigmine reversal dosing is determined based on the degree of blockade observed through quantitative TOF monitoring, and extubation is performed when the measured TOF ratio is ≥ 0.90.
  Interventions: Device: Train of four monitoring device intraoperative; Drug: Neostigmine; Procedure: Air chalenge prior to extubation; Device: Train of Four monitoring device in recovery room

INTERVENTIONS:
Device: Train of four monitoring device intraoperative — Only group B will receive reversal strategy based on the presence of TOF monitoring device prior to extubation. If they meet the criteria, patients will then be extubated.
  Arms: Clinical extubation strategy with TOF monitoring
Drug: Neostigmine — For subjects in Group A, the first researcher calculated the time of the last administration of the muscle relaxant and the subject's spontaneous breathing efforts. Neostigmine was administered based on the reversal protocol. For subjects in the TOF monitoring group (Group B), the first researcher attached the TOF monitoring device. After it was attached and turned on, TOF stimulation was provided without calibration, with a stimulation intensity of 50 mA. Measurements were taken in a 12-second cycle mode. Neostigmine was administered according to the measured TOF value at the start of skin/muscle closure as the protocol.
  Other Names: Neuromuscular blockade reversal
Procedure: Air chalenge prior to extubation — After surgery was completed and the TOF ratio was ≥ 0.90, the TOF device was removed, and extubation was performed in Group B. In Group A, after a minimum of 15 minutes following reversal, patients received only ambient air without supplemental O2. Extubation was performed if the patient could maintain an SpO2 > 95% for a minimum of 3 minutes. If within 15 minutes after reversal the patient did not meet the extubation criteria, the degree of blockade was reassessed, and a repeat dose of neostigmine and atropine was administered as needed. If there was suspicion of opioid-induced hypoventilation, naloxone was administered at 0.4-0.8 mcg intravenously.If the patient was unable to maintain oxygen saturation for the 3-minute duration, oxygen supplementation was reinstated, the degree of blockade was reassessed, and a repeat dose of neostigmine and atropine was administered as needed.
Device: Train of Four monitoring device in recovery room — Upon arrival in the recovery room, all subjects were fitted with SpO2, EKG, NIBP monitors, and the TOF monitoring device. TOF values were measured by a second researcher who was unaware of the type of intervention. Measurements were taken twice sequential

SUMMARY:
Patients undergoing general anesthesia will have an endotracheal tube inserted. Adequate muscle strength recovery in the recovery room is crucial to ensure before extubation. One of the criteria we use to determine the recovery of muscle strength post-use of muscle relaxants in conditions without specific monitoring devices is the ability to maintain body oxygen levels without oxygen assistance for 3 minutes. This study aims to determine the muscle strength value in the recovery room using extubation strategies without muscle strength monitoring compared to extubation strategies with muscle strength monitoring.

DETAILED DESCRIPTION:
The availability of Train-of-Four (TOF) monitoring devices is not yet widespread in some clinical practices. Practitioners are also often unaware of the high incidence of residual paralysis and the associated risks in their daily practice. However, residual paralysis increases the occurrence of airway obstruction, hypoxemia, and postoperative pulmonary complications. Therefore, clinical parameters for extubation criteria must ensure the absence of residual paralysis.

Administering oxygen in the ambient air can identify hypoventilation conditions. Therefore, patients who can maintain oxygen saturation levels > 95% can be considered not experiencing hypoventilation. The author aims to validate ventilation adequacy as an additional clinical parameter for extubation criteria without TOF monitoring to ensure the absence of residual paralysis in the recovery room.

This study is planned using a randomized controlled trial method with observer blinding. The study consists of 3 comparisons based on the type of volatile anesthetic gas agent and neuromuscular blockade agent. This research will involve 240 subjects aged 18-60 years undergoing elective surgery under intubation general anesthesia. Subjects will be divided into two parallel treatment groups randomly stratified by the type of surgery to observe the incidence rate of residual paralysis in the recovery room. Group A will receive extubation strategy without additional oxygen supplementation, while Group B will use extubation strategy with quantitative TOF monitoring.

Group A will receive optimal reversal strategy using neostigmine based on clinical criteria such as tidal volume adequacy and the time of last administration of the neuromuscular blockade agent. Then, patients will be assessed 15 minutes after reversal for the ability to maintain oxygen saturation levels > 95% without oxygen supplementation. If they meet these criteria, patients will then be extubated. Group B will receive optimal reversal strategy using neostigmine based on TOF values. If the measured TOF value is ≥0.90, patients can be extubated while awake. Upon arrival in the recovery room, the TOF values of both groups will be measured and compared as the outcome of this study.

The results of this study are expected to provide recommendations for extubation strategies based on clinical parameters to clinicians with limited access to TOF monitoring devices. With the implementation of this change in extubation strategy, unexpected post-anesthesia events may be reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery
2. Adult patiens aged 18-60 years
3. ASA physical status I-II
4. Not receiving oxygen supplementation during pre-operative care

Exclusion Criteria:

1. History of hypersensitivy or allergy to neostigmine, muscular blockade agents, or anesthetic agents given
2. Head or neck surgery
3. Inability to access the ulnar nerve for TOF measurement device placement
4. History of lung diseases such asthma, COPD, or pleural effusion
5. Hepatic impairment with liver enzyme values > 50% of the normal range
6. Renal insufficiency (serum creatinine > 1.8 mg/dl) or kidney failure
7. Patients with neuromuscular diseases
8. Body mass index (BMI) > 35 kg/m2
9. Consumption of medications that affect neuromuscular transmission such as aminoglycoside, polymyxin, lincomycin, clindamycin, and tetracycline; local anesthetic agent, procainamide, quinidine, lithium, magnesium sulfate, furosemide, cyclosporine, dantrolene, anti-estrogens, anticonvulsant, calcium, steroid, and azathioprine.
10. Patients with contraindications to neostigmine or atropine sulfate
11. Planned post-operative intensive care unit treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Residual paralysis in recovery room | Up to 30 minutes in recovering room
  Residual paralysis in the recovery room was defined as a condition with a measured TOF ratio < 0.90 upon arrival in the recovery room. TOF values were measured by a second researcher who was unaware of the type of intervention. Measurements were taken twice sequentially with a 12-second interval. The value used was the average of these two measurements. However, if the values differed by >10%, two more measurements were taken using the same method. The value used was the average of the two closest values out of the four measurements.

SECONDARY OUTCOMES:
Adverse events | Up to 30 minutes in recovering room
  Any adverse respiratory events such as upper airway obstruction, hypoxemia, respiratory distress, and reintubation; Severe allergic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Sardjito General Hospital, Yogyakarta, Indonesia